CLINICAL TRIAL: NCT03875768
Title: Using Digital Health to Improve Diet Quality Among Adults at Risk for Cardiovascular Disease
Brief Title: Nourish: A Digital Health Program to Promote the DASH Eating Plan Among Adults With High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00101689
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-03

CONDITIONS: Hypertension; Health Behavior
Keywords: Blood pressure; Hypertension; DASH; Nutrition; Dietary change; Mobile health; Digital health; E-health
MeSH Terms: conditions — Hypertension; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will track their daily dietary intake for six months using an app and will receive automated feedback daily via text message based on DASH nutrients. Participants in-need of coaching based on their adherence to the key nutrients in the DASH dietary pattern or engagement in the intervention will receive responsive digital coaching from Nourish registered dietitians.
  Interventions: Behavioral: Tracking plus coaching
- Control (No Intervention): Participants will receive information about the DASH dietary pattern and will track their daily dietary intake using an app for six months.

INTERVENTIONS:
Behavioral: Tracking plus coaching — Participants will track their nutrition intake every day for six months using a study app and receive tailored feedback via text message based on their nutritional intake and adherence to the DASH dietary pattern. If necessary, they will receive responsive coaching from a Nourish registered dietitian in order to increase adherence to the DASH dietary pattern and their engagement with the intervention.
  Arms: Intervention

SUMMARY:
The goal of Nourish is to help adults with high blood pressure enjoy an eating pattern called DASH (Dietary Approaches to Stop Hypertension) to lower blood pressure and improve health. Nourish will use a mobile app and information about DASH to help study participants follow the DASH dietary plan by tracking what they eat and drink every day. The primary outcome of the study is 6-month change in following the DASH eating plan, as measured by 24-hour dietary recalls. The secondary outcome is change in blood pressure. Study participation will last one year.

DETAILED DESCRIPTION:
Over 100 million Americans suffer from high blood pressure and are at increased risk for cardiovascular disease. Evidence supports the DASH (Dietary Approaches to Stop Hypertension) dietary pattern to reduce blood pressure. DASH is rich in fruits and vegetables, legumes, lean protein, and low-fat dairy, and reduced in red meats, sweets and processed foods. The Nourish trial will look at the effect of the intervention on changes in dietary quality and blood pressure among men and women with high blood pressure. Participants who join Nourish will be asked to track what they eat and drink every day through a smartphone app and to participate in online study visits. Some participants will also receive additional support from a registered dietitian. We are doing this study to understand how technology can help adults with high blood pressure follow a heart-healthy eating plan to improve their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure of 120-159 mmHg or diastolic blood pressure of 80-99 mmHg, whether or not taking blood pressure medications.
* BMI ≥ 18.5 kg/m2
* Smartphone with a data plan
* Willing to receive daily text messages
* Valid email address
* Willing and able to participate in online study videoconferencing visits (Zoom)
* Lives in the U.S.
* Reads and writes in English

Exclusion Criteria:

* Participating in another related research study
* Cardiovascular disease event (e.g. stroke, myocardial infarction) in prior 6 months
* Bariatric surgery in the last 12 months or planned during the study period
* Active cancer
* Recent hospitalization due to psychiatric condition or event
* Pregnancy- current or planned during the study period
* Documented dementia
* Lives with someone else participating in the Nourish study

To learn more about the study and to see if eligible to participate, visit www.nourishstudy.org

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary G. Bennett, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention - Tracking Plus Coaching: Participants will track their daily dietary intake for six months using an app and will receive automated feedback daily via text message based on DASH nutrients. Participants in-need of coaching based on their adherence to the key nutrients in the DASH dietary pattern or engagement in the intervention will receive responsive digital coaching from Nourish registered dietitians.
  Tracking plus coaching: Participants will track their nutrition intake every day for six months using a study app and receive tailored feedback via text message based on their nutritional intake and adherence to the DASH dietary pattern. If necessary, they will receive responsive coaching from a Nourish registered dietitian in order to increase adherence to the DASH dietary pattern and their engagement with the intervention.
- Attention Control: Participants will receive information about the DASH dietary pattern and will track their daily dietary intake using an app for six months.
Period: Overall Study
Arm/Group | Intervention - Tracking Plus Coaching | Attention Control
Started | 150 | 151
Completed | 102 | 105
Not Completed | 48 | 46
Not completed — Lost to Follow-up | 16 | 13
Not completed — Withdrawal by Subject | 10 | 21
Not completed — Did not complete assessment | 21 | 12
Not completed — Became ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - Tracking Plus Coaching | Attention Control | Total
Number analyzed (Participants) | 150 | 151 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (13.1) | 53.4 (13.6) | 54.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 95 | 196
  Male | 49 | 56 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 139 | 140 | 279
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 53 | 100
  White | 89 | 83 | 172
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 150 | 151 | 301

OUTCOME MEASURES:

1. Primary Outcome: Change in Dietary Intake as Measured by Dietary Approaches to Stop Hypertension (DASH) Score
Description: Participants entered their dietary intake online via the National Cancer Institute's Automated Self-Administered 24-hour (ASA24) Dietary Assessment tool to record 2 separate 24-hour dietary recalls (1 weekday and 1 weekend day). DASH dietary nutrients are then converted into a score using the method described in Mellen et al (2008). Scores ranged from 0 to 9 where a higher score indicates better adherence to the DASH dietary pattern. Change in DASH score = 6-month DASH score - Baseline DASH score.
Time Frame: Baseline and 6 months
Population: Participants who completed the baseline and 6-month dietary recalls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention - Tracking Plus Coaching | Attention Control
Number analyzed (Participants) | 102 | 105
score on a scale | 0.3 (1.7) | 0.3 (1.8)
Statistical Analysis 1: Comparison: Intervention - Tracking Plus Coaching vs Attention Control; The expected effect size is 0.5. The investigators hypothesize that the intervention will lead to an increase in average DASH score of 2 units. The investigators used a standard deviation for 2 units for both intervention and attention control groups since higher variability may be observed with a bigger sample size than the pilot study; Test type: Superiority; p = 0.89, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Results presented are unadjusted; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.44 to 0.50], Standard Deviation 1.72

2. Secondary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure measured in millimeters of mercury (mmHg) using the upper arm three times at 1-minute intervals after 5 minutes of quiet sitting. Blood pressure was measured 3 times at 1 minute intervals. The final 2 measurements were averaged together for analysis. Change in systolic blood pressure = 6-month systolic blood pressure - Baseline systolic blood pressure.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention - Tracking Plus Coaching | Attention Control
Number analyzed (Participants) | 122 | 113
mmHg | -5.5 (13.0) | -3.5 (12.9)
Statistical Analysis 1: Comparison: Intervention - Tracking Plus Coaching vs Attention Control; The expected effect size for change in systolic blood pressure (SBP) between intervention and control group is 0.6 based on the pilot study. With a 90% power and a type I error rate (alpha) of .01, the investigators can detect the expected effect size with the proposed sample size of 121 per study arm; Test type: Superiority; p = 0.26, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Results presented are unadjusted; Mean Difference (Net) = -1.9, 95% CI 2-sided [-5.3 to 1.4], Standard Deviation 13.0

3. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Diastolic blood pressure measured in millimeters of mercury (mmHg) using the upper arm three times at 1-minute intervals after 5 minutes of quiet sitting. Blood pressure was measured 3 times at 1 minute intervals. The final 2 measurements were averaged together for analysis. Change in diastolic blood pressure = 6-month diastolic blood pressure - Baseline diastolic blood pressure.
Time Frame: Baseline and 6 months
Population: Participants who completed the blood pressure assessment protocol.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention - Tracking Plus Coaching | Attention Control
Number analyzed (Participants) | 122 | 113
mmHg | -3.0 (8.6) | -2.1 (7.9)
Statistical Analysis 1: Comparison: Intervention - Tracking Plus Coaching vs Attention Control; The expected effect size for change in diastolic blood pressure (DBP) between intervention and control group is 0.75 based on the pilot study. With a 90% power and a type I error rate (alpha) of .01, the investigators can detect the expected effect size with the proposed sample size of 121 per study arm; Test type: Superiority; p = 0.39, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Results presented are unadjusted; Mean Difference (Net) = -0.9, 95% CI 2-sided [-3.1 to 1.2], Standard Deviation 8.3

ADVERSE EVENTS:
Time Frame: Randomization through 12 months (final endpoint of trial)
Arm/Group | Intervention - Tracking Plus Coaching | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/151
Serious Adverse Events (participants affected / at risk) | 6/150 | 15/151
Other Adverse Events (participants affected / at risk) | 28/150 | 21/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention - Tracking Plus Coaching (N=150) | Attention Control (N=151)
Cardiovascular issues (pacemaker, MI, afib, etc.) (Cardiac disorders) | 2 | 2
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
COPD related (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Mental health issues (Psychiatric disorders) | 1 | 0
Broken limbs/accidents (Injury, poisoning and procedural complications) | 2 | 3
Arthritis (Immune system disorders) | 0 | 1
Detached retina (Eye disorders) | 0 | 1
Choking (Gastrointestinal disorders) | 0 | 1
Urological issues (Renal and urinary disorders) | 0 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 1
Breast reconstructive surgery (Reproductive system and breast disorders) | 1 | 0
Parkinsons (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention - Tracking Plus Coaching (N=150) | Attention Control (N=151)
Issues with eyes (Eye disorders) | 1 | 0
Sinus/respiratory issues (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Various medical procedures (Surgical and medical procedures) | 4 | 5
GI issues (Gastrointestinal disorders) | 5 | 2
Mental health challenges (Psychiatric disorders) | 1 | 0
Fractured bones/torn ligaments (Musculoskeletal and connective tissue disorders) | 2 | 2
Heart rate/BP/ afib (Cardiac disorders) | 5 | 6
Immune-related issues (Immune system disorders) | 2 | 0
Infections from ticks (Infections and infestations) | 1 | 1
Kidney related issues (Renal and urinary disorders) | 2 | 0
Cancer related issues (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Accidents (Injury, poisoning and procedural complications) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT03875768/Prot_SAP_ICF_001.pdf